CLINICAL TRIAL: NCT04310631
Title: Optical Coherence Tomography Angiography Findings After Intravitreal Ranibizumab in Patients With Coats Disease
Brief Title: Evaluation of Retinal and Vascular Features in Coats Disease After Intravitreal Injections of Ranibizumab
Status: Completed | Type: Observational
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Gilda Cennamo, Principal Investigator, Federico II University
Other Study IDs: PT1003/20
Record Dates: First submitted 2020-03-10; First posted 2020-03-17 (Actual); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: Coats Disease
MeSH Terms: conditions — Retinal Telangiectasis | interventions — Ranibizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Ranibizumab Injection — Ranibizumab Injection (0.5 mg/0.05 ml): Three monthly intravitreal injections

SUMMARY:
This study evaluates the retinal and vascular features in patients affected by Coats disease under the effects of Ranibizumab intravitreal injections using optical coherence tomography and optical coherence tomography angiography

DETAILED DESCRIPTION:
Coats disease is an idiopathic retinal vascular disorder, occurs in young males, and is characterized by retinal telangiactasias, numerous yellowish exudates in the subretinal space, macular edema, hemorrhages and, in advanced end-stage, by exudative retinal detachment.

Ranibizumab is a vascular endothelial growth factor antagonist represent an efficacy treatment acting on vascular hyperpermeability. The optical coherence tomography and optical coherence tomography angiography represent novel and non-invasive diagnostic techniques that allow a detailed analysis of retinal and vascular features. The study evaluates the changes in optical coherence tomography and optical coherence tomography angiography parameters at baseline and after three monthly injections of Ranibizumab in Coats disease.

ELIGIBILITY:
Inclusion Criteria:

* age older than 18 years
* diagnosis of Coats disease
* treatment-naïve with Ranibizumab
* absence of other vitreoretinal and vascular retinal diseases
* absence of diabetes

Exclusion Criteria:

* age younger than 18 years
* No diagnosis of Coats disease
* previous treatments with Ranibizumab
* presence of vitreoretinal and vascular retinal diseases
* presence of diabetes

Ages: 19 Years to 30 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Study Population: The participans were older than 18 years with diagnosis of Coats disease. They did not present other ophthalmological diseases.
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Study of retinal and vascular features in Coats disease after intravitreal injections of Ranibizumab | Three months
  The effectiveness of Ranibizumab injections for treating Coats disease using optical coherence tomography (OCT).
  The parameters analyzed by OCT were:
  Central Macular Thickness (micron), Subfoveal Choroidal Thickness (micron)
Study of retinal and vascular features in Coats disease after intravitreal injections of Ranibizumab | Three months
  The effectiveness of Ranibizumab injections for treating Coats disease using optical coherence tomography angiography (OCTA)
  The parameters analyzed by OCTA were:
  retinal vessel density (%), choriocapillaris vessel density (%)

CONTACTS AND LOCATIONS:
Overall Officials: Gilda Cennamo, Principal Investigator — Federico II University; Daniela Montorio, Study Director — Federico II University
Locations (1):
- University of Naples "Federico II", Naples, Italy